CLINICAL TRIAL: NCT07180381
Title: Sequential Imaging of Suspicion of Prostate Cancer Reducing Overdiagnosis and Unnecessary Biopsy With Timely Diagnosis of Significant Cancer
Acronym: SPROUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Harm H.E. Van Melick, MD PhD, St. Antonius Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL-005445
Record Dates: First submitted 2025-07-16; First posted 2025-09-18 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Participants will not undergo immediate prostate biopsy but will be monitored with PSA testing every six months and prostate MRI annually.
  Interventions: Other: PSA and MRI-monitoring

INTERVENTIONS:
Other: PSA and MRI-monitoring — Men with PI-RADS 3 or 4 lesions and a PSA density ≤ 0.15 ng/mL² are actively monitored with PSA testing every six months and MRI annually, instead of undergoing immediate prostate biopsy.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of a novel diagnostic strategy for prostate cancer, in which men with a moderate risk of prostate cancer are monitored using PSA and MRI instead of immediate biopsy,.

The main questions it aims to answer are:

* Is it safe to delay biopsy, making sure that clinical significant prostate cancers are not often missed?
* Does it reduce unnecessary biopsies and overtreatment?

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy > 10 years
* initial PSA < 20 ng/ml
* No signs of extracapsular disease on digital rectal examination
* Intermediate-risk category for suspicion of prostate cancer determined by MRI results and PSA density (PSAD): PI-RADS 3 or PI-RADS 4 with PSAD =< 0.15
* Mentally competent and able to comprehend the potential benefits and burdens of the study
* Willing to undergo the follow-up protocol for a maximum of four years
* written and signed informed consent

Exclusion Criteria:

* Men who have previously undergone a prostate biopsy
* Men who have a prior PCa diagnosis
* using any (anti-)hormonal therapy, including 5-alpha-reductase inhibitors
* Proven germline mutation for PCa (for example: BRCA1; BRCA2)
* Secondary malignancy, besides basal cell carcinoma of the skin, for which the potential participant is receiving active treatment at the time of inclusion.
* severe claustrofobia or other conditions that make (repeat) MRI unsuitable (e.g., metal implants, pacemakers)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Proportion clinically significant prostate cancer missed during follow up | 48 months
  Detection percentage of International Society of Urological Pathology Grade Group (ISUP GG)≥ 2 prostate cancer (= clinically significant prostate cancer) during 48 months of follow up compared with the percentage of total ISUP GG≥ 2 during the study, including any findings from end of study biopsies.
  ISUP grade groups range from 1 to 5, and a ISUP GG≥ 2 is defined as clinically significant prostate cancer.
Number of clinically insignificant prostate cancer detected | 48 months
  Detection of clinically insignificant prostate cancer (International Society of Urological Pathology Grade Group (ISUP GG) 1) during the 48 months of follow up compared to the total ISUP GG 1 including end of study biopsies.
Number of negative biopsies | 48 months
  Number of participants with negative biopsy results during the study including findings from the end of study biopsies.

SECONDARY OUTCOMES:
Grade shifts | 48 months
  Progression rates of intermediate- to high-risk group during monitoring, rates of downgrading from intermediate risk to low risk
Detection of very high risk prostate cancer | 48 months
  Detection of very high risk prostate cancer (ISUP GG ≥ 3) during the study, including end of study biopsies.
Health-related quality of life (EPIC-26 score) | 48 months
  Change in health-related quality of life as measured by the Expanded Prostate Cancer Index Composite (EPIC-26), a validated questionnaire with subscales ranging from 0 to 100. Higher scores indicate better function and less symptom burden. Although the diagnosis of prostate cancer is not confirmed, this is the best validated and suitable questionnaire. Participants will be asked to fill in the questionnaire once a year.
Estimated average cost per patient during 48-month follow-up | 48 months
  Mean cost per participant over 48 months, including diagnostics (e.g. MRI, biopsies), consultations, and treatments, based on predefined unit costs and healthcare utilization.
Anxiety symptomes (STAI-6 score) | 48 months
  Change in anxiety levels as measured by the 6-item short form of the State-Trait Anxiety Inventory (STAI-6), with scores ranging from 20 to 80. Higher scores indicate greater anxiety. Participants will be asked to fill in the questionnaire once a year.

CONTACTS AND LOCATIONS:
Locations (7):
- Netherlands (7):
  - Treant, Emmen, Drenthe
  - Andros Clinics, Arnhem, Gelderland
  - Radboud University Medical Centre, Nijmegen, Gelderland
  - Canisius Wilhelmina Hospital, Nijmegen, Gelderland
  - Antoni van Leeuwenhoek Hospital, Amsterdam, North Holland
  - Maasstad Hospital, Rotterdam, South Holland
  - St Antonius Hospital, Nieuwegein, Utrecht

IPD SHARING:
Plan to Share IPD: No